CLINICAL TRIAL: NCT07273253
Title: Multimodal Intervention for Older Adults Residing in Temporary Housing After an Earthquake: A Randomized Controlled Study
Brief Title: Multimodal Intervention for Older Adults After an Earthquake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Yusuf Şinasi Kirmaci, Assistant Professor, PhD, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EARTHQUAKE_GERIARTRIC_1
Record Dates: First submitted 2025-11-19; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Frailty at Older Adults; Post-Traumatic Stress Disorder in Old Age; Depression in Adults; Malnutrition Elderly; Falls (Accidents) in Old Age
Keywords: Older adults,; Earthquake survivors,; Temporary housing,; Container housing,; Health management program,; Rehabilitation,; Exercise,; Balance,; Physical activity; Nutrition education; Post-disaster; Frailty; Kahramanmaras
MeSH Terms: conditions — Motor Activity; Frailty

STUDY DESIGN:
Intervention Model Description: study and control groups
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Individuals over the age of 65 who experienced the earthquake
  Interventions: Other: Multimodal intervention
- Control Group (No Intervention): Individuals over the age of 65 who experienced the earthquake

INTERVENTIONS:
Other: Multimodal intervention — Pre-earthquake and post-earthquake health problems were identified, and general health status was assessed using a holistic approach. A health management plan was developed to address changing health priorities, and this plan was implemented by the participants under the supervision and consultancy of the researchers. A three-month health management plan and observation were conducted to determine the impact of the health management plan and recommendations on quality of life. Participants' general health status was reassessed at the end of the study.
  Arms: Study Group

SUMMARY:
This randomized controlled study was conducted among older adults (≥65 years) living in temporary container housing in Kahramanmaraş after the February 2023 earthquakes. A total of 60 participants meeting inclusion criteria were recruited and randomized into two groups: an intervention group (n=30) and a control group (n=30). Randomization was performed using a sealed envelope method following minimization based on frailty scores (Edmonton Frailty Scale ≥4).

The intervention group received a 12-week health management program designed with a holistic approach, addressing physical, mental, and nutritional health needs. Individualized exercise prescriptions (balance, strength, range of motion, posture correction), lifestyle counseling, nutrition education, and medication use training were provided under professional supervision. The control group received no active intervention and only underwent assessments at baseline and at the end of the study.

Measurements were performed at baseline and after 12 weeks. Primary assessments included frailty status (Edmonton Frailty Scale), balance and mobility (Berg Balance Scale, Timed Up and Go Test, Functional Reach Test, Gyko postural sway analysis), physical activity level (PASE questionnaire), physical performance (Short Physical Performance Battery), muscle strength (hand dynamometer, pinch meter, digital force measurement), posture (PostureScreen app), and nutritional status (Mini Nutritional Assessment, anthropometric measures). Cognitive and mental health were evaluated using the Mini-Mental State Examination (MMSE) and the Geriatric Anxiety Scale. Quality of life was assessed with the Nottingham Health Profile.

The study aims to determine whether a structured, holistic health management plan can improve balance, physical activity, and overall health outcomes compared with control in older adults living in post-disaster temporary housing. Findings are expected to inform rehabilitation and preventive health strategies for vulnerable elderly populations in disaster settings.

DETAILED DESCRIPTION:
This randomized controlled trial was designed to address the health priorities of older adults (≥65 years) living in temporary container housing following the devastating Kahramanmaraş earthquakes in February 2023. Recognizing the unique vulnerabilities of elderly individuals in post-disaster environments - such as frailty, physical inactivity, limited access to care, and psychosocial distress - the study implemented a multidisciplinary, holistic intervention targeting their comprehensive health needs.

Participants were allocated into two groups (intervention and control) based on frailty stratification using the Edmonton Frailty Scale and randomized using a sealed-envelope method. The intervention group received a 12-week individualized health management program, tailored to physical, mental, and nutritional domains. The program was developed and delivered by a multidisciplinary team including physiotherapists, geriatric nurses, nutritionists, and mental health professionals.

The intervention included:

Physical health sessions: individualized exercise plans for posture correction, mobility, strength, and balance.

Nutritional counseling: personalized dietary education based on individual risk factors and nutritional deficiencies.

Mental health support: education on coping mechanisms, peer group interaction, and anxiety-reducing strategies.

Medication education: safe drug use training, including awareness of polypharmacy and drug-food interactions.

All sessions were conducted in person within the container housing area, considering participants' mobility limitations. Adherence was monitored throughout the study. The control group underwent only baseline and 12-week follow-up assessments and received no active intervention during the trial period.

This trial aims to demonstrate the feasibility and effectiveness of a holistic health model in disaster-stricken elderly populations. The approach moves beyond disease management, incorporating lifestyle reorganization and psychosocial support. The findings are intended to contribute to the creation of post-disaster rehabilitation guidelines and policies for geriatric populations in similar emergency settings.

ELIGIBILITY:
Inclusion Criteria:

* Living in a container city,
* Scoring 4 or below on the vulnerability scale,
* Being an earthquake victim,
* Being able to understand verbal commands and being over 65 years of age,
* Being able to speak and understand Turkish,
* Volunteering to participate in the research.

Exclusion Criteria:

* Not being an earthquake victim,
* Not living in a container,
* Being under 65 years of age,
* Not knowing or understanding Turkish,
* Not wanting to participate in the study,
* Not being able to understand verbal commands,
* Having received any psychological diagnosis,
* Having undergone any surgery within the last 6 months,
* Scoring 5 or above on the frailty scale.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Daily Living and Instrumental Activities Scale | 1.week and 12.week intervention
  The instrumental activities of daily living scale consists of eight items measuring an individual's ability to make phone calls, shop, prepare meals, do housework, do laundry, use transportation, take their own medication, and manage their finances. A participant can receive a minimum of 8 and a maximum of 24 points. A score range of 0-8 indicates that the participant is dependent in instrumental activities of daily living, a score range of 9-16 indicates that the participant is semi-dependent, and a score range of 17-24 indicates that the participant is independent. A higher scale score indicates a higher degree of independence.
Physical Activity Scale For The Elderly (PASE) | 1.week and 12.week intervention
  The PASE examines the intensity, frequency, and duration of physical activities such as walking; light, moderate, and strenuous sports and recreational activities; muscle-strengthening and endurance exercises; work-related activities, including walking and standing; lawn and garden care; caregiving; home repairs; and assesses both strenuous and light household activities performed by participants in the past week. the overall PASE score ranges from 0 to 400 or more, with higher scores indicating better physical activity levels.
Posture Screen mobile app | 1.week and 12.week intervention
  The Posture Screen mobile app allows you to quickly capture posture images using photography in frontal and lateral stances. This app identifies postural deviations.
The Short Physical Performance Battery | 1.week and 12.week intervention
  The Short Physical Performance Battery (SPPB) is widely used to assess the physical and functional health of elderly people living in the community (20). The SPPB consists of three objective tests that assess lower body function: a 4-meter walk, a chair rise, and a standing balance test. A 5-level summary score (0-4) is assigned to each test. A score of zero indicates "failure to perform." Participants included in the "failure to perform" category were: 1. Those who attempted but were unable to perform the activity, 2. Those who felt unsafe due to the interviewer or the subject, and 3. Those who were unable to perform the activity due to other health reasons. The scores 1-4 obtained by the subjects indicate the progressive performance required to complete the test according to the times specified below.
Muscle Strength Measurement | 1.week and 12.week intervention
  It will be evaluated by isometric strength measurement of bilateral serratus anterior, trapezius, deltoid, supraspinatus, teres minor, biceps brachii muscles of the upper extremity and bilateral iliopsoas, gluteus medius, gluteus maximus, hamstring, quadriceps femoris, tibialis anterior muscles of the lower extremity with a digital muscle strength measurement device (KFORCE KINVENT digital muscle strength measurement device).
Grip strength measurement | 1.week and 12.week intervention
  Jamar hand dynanometer (Baseline®) (Svens B, 2005) and PinchMetre Pinch Meter (Baseline Mechanical Pinch Gauge With Case, Blue, 30 Lb) (Dukelow NJ, 1996) will be used for grip strength measurement.
Timed Up and Go Test (TWAT) | 1.week and 12.week intervention
  Timed Up and Go Test (TWAT) is a reliable test that measures walking speed, postural control, functional mobility, and balance. TWAT is a clinical measure that is easy to administer to older adults and indicates the risk of falls.
Postural Sway and Balance Assessment | 1.week and 12.week intervention
  Postural Sway and Balance Assessment with Gyko: This device determines three main measures of body sway: sway length and area, sway progression rate, and sway frequency. Postural analysis is objectively performed through biomechanical movement analysis, with changes in minimal postural adjustments. This device measures postural sway, sway length, sway duration, and frequency. Used to assess and measure individuals' balance in various situations and/or on various surfaces, Gyko measures this by detecting postural sway in forward-backward, medial-lateral directions, and changes and imbalances within the support surface. By determining the main directions and amplitude of trunk movement, this device records the movement.
Nutritional evaluation | 1.week and 12.week intervention
  Nutritional evaluation; eating habits, body mass index, waist/hip ratio, and fat type will be determined.
Food Consumption Frequency | 1.week and 12.week intervention
  Food Consumption Frequency Form: This form will be used to determine the frequency and quantity of food groups or foods consumed. Consumption frequency is given by day, month, or week. Food consumption frequency provides information about an individual's dietary pattern. It is a frequently used method for assessing the relationship between nutrition and health. The food consumption frequency form can be prepared differently depending on the purpose of the person preparing it. Foods are listed as a single statement or by classification (full-fat, low-fat, or fat-free). The food consumption frequency form used in the study includes a total of 18 food items. The food groups are milk and dairy products, meat, eggs, legumes, vegetables and fruits, grains, fats and sweets, and beverages. Participants will be asked how often they consume the food (1-2 times a day, 1-3 times a week, 4-6 times a week, once every 15 days, once a month, never) to determine their daily energy and nutrient intake.
Body Mass Index | 1.week and 12.week intervention
  Body Mass Index: Individuals' body weights will be measured using a scale with a capacity of at least 100 g and 150 kg, and their heights will be measured using a non-flexible tape measure, held in the Frankfurt plane, with shoes and feet together and not fixed to a wall. BMI values will be calculated by dividing individuals' body weight (kg) by the square of their height (kg/m2), and they will be classified according to the WHO BMI classification.
Waist and hip circumference | 1.week and 12.week intervention
  Waist circumference will be measured with a 0.1 cm precision, non-flexible tape measure, with the individual standing, arms relaxed, feet together, and the midpoint between the lower rib and the groin without applying pressure.
  Hip circumference will be measured with the individual standing upright, with the researcher holding the tape measure parallel to the floor, at the skin level of the trochanterion points of the femur. The measurement will be taken with the tape measure parallel to the floor and taut. The measurement will be recorded in millimeters.
Waist/Hip Ratio | 1.week and 12.week intervention
  Waist/Hip Ratio: According to the World Health Organization, when determining obesity, body mass index, waist circumference, and waist-hip ratio methods are used, a ratio of 0.85 or higher in women and 0.90 or higher in men will be considered obese.
Nutritional Assessment | 1.week and 12.week intervention
  Nutritional Assessment; Mini Nutrition Test (MNA), whose Turkish validity and reliability study was conducted by Sarıkaya (2013), is one of the most frequently used tests to screen for nutritional status and indicate the risk of malnutrition in older adults. The MNA test consists of 18 questions: 6 screening and 12 assessment questions. Fifteen of these questions are verbal questions and three are anthropometric measurements. The nutritional score is evaluated out of 30 points. A score of 12 or higher out of 14 in the six-question preliminary questioning section is considered normal, and the test is terminated. Individuals who score 11 or less in this section continue with the remaining 12 questions. A total score of <17 indicates definite malnutrition, 17-23 indicates risk of malnutrition, and 23.5-30 indicates normal nutritional status.
Mental State Examination | 1.week and 12.week intervention
  Mini Mental State Examination: The Mini Mental State Examination (MMSE), which is highly suitable for screening cognitive function in the elderly and assesses cognitive functions in five separate areas (orientation, registration, attention and calculation, recall, and language), is frequently used. A score below 24 on the MMSE indicates dementia, 24-26 indicates mild cognitive impairment, and 26 or above indicates normal cognitive function.
Geriatric Anxiety | 1.week and 12.week intervention
  Geriatric Anxiety Scale (GAS) aims to measure anxiety symptoms in the elderly dimensionally. The scale's fundamental psychometric property is its ability to distinguish between those with and without anxiety and those with and without generalized anxiety disorder. The cut-off point for generalized anxiety disorder is set at 10/11. Accordingly, the scale is structured as "anxiety symptoms and generalized anxiety disorder > 10; anxiety symptoms only < 10." The 20-item scale, scored on two dimensions: "agree" and "disagree," contains no reverse-coded items. Therefore, "agree" is assigned 1 point and "disagree." Therefore, scale scores can range from 0 to 20.
Health Care Assessment | 1.week and 12.week intervention
  Health Care Assessment; Nottingham Health Profile (NSP), available in Turkish, is a measurement tool that assesses individuals' health problems and how these problems impact their daily activities. It is used to assess the quality of life of older adults. The NSP consists of 38 items across six dimensions. The subdimensions are: energy level (ES), emotional reactions (ER), physical activity (PA), pain (A), sleep (U), and social isolation (SI). It is a general health questionnaire consisting of 38 items and six subparameters. Answers to the questions are given as "yes" or "no" based on the current situation.

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Şinasi KIRMACI, Assist.Prof, Principal Investigator — Kahramanmaras Sutcü Imam University
Locations (1):
- Kahramanmaras Sutcu İmam University, Kahramanmaraş, Turkey (Türkiye)